CLINICAL TRIAL: NCT02758860
Title: Predictive Value of the Diverticular Inflammation and Complication Assessment (DICA) Endoscopic Classification on the Outcome of the Diverticular Disease of the Colon: a Prospective, Multicenter, International Study.
Brief Title: Predictive Value of DICA in the Diverticular Disease of the Colon
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Erasmo Spaziani, Professor, University of Roma La Sapienza
Other Study IDs: DICA Trial
Record Dates: First submitted 2016-04-23; First posted 2016-05-03 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Colonic Diverticula
Keywords: Colonoscopy; Diverticular disease of the colon; Classification
MeSH Terms: conditions — Diverticulum, Colon | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Colonoscopy — Patients will be submitted to diagnostic colonoscopy

SUMMARY:
The Diverticular Inflammation and Complication Assessment (DICA) is an endoscopic classification for diverticulosis and diverticular disease of the colon.

The aim of the study is to show that DICA classification is a valid parameter to predict the risk of acute diverticulitis occurrence/recurrence and the need of surgery in patients suffering from diverticulosis/diverticular disease of the colon.

DETAILED DESCRIPTION:
The Diverticular Inflammation and Complication Assessment (DICA) endoscopic classification has been recently developed for patients suffering from diverticulosis and diverticular disease.

A recent multicentre, international, retrospective study found that DICA classification has a significant predictive value on the outcome of the disease in terms of acute diverticulitis occurrence/recurrence and surgery occurrence.

The aim of the present study is to confirm the above mentioned results propectively Several centers, worldwide distributed, will be involved. A minimum of 281 patients will be required for the study. This calculation will be based on the assumption that a continuity-corrected chi-square test with a type I error of 0.05 and a type II error of 0.20 will be expected to detect a difference between a 4.3% prevalence of diverticulitis in patients with diverticulosis and 8.6% in DICA I patients.

Only patients at the first endoscopic diagnosis of diverticulosis/diverticular disease will be enrolled. For each patient, we recorded: age; severity of DICA score; severity of symptoms at entry and during the follow-up; C-reactive protein (CRP) and fecal calprotectin test at the time of diagnosis and during the follow-up (CRP only for DICA 2 and 3 patients); comorbidities (if any); concomitant therapies (if any); therapy taken during the follow-up to maintain remission (if any); months of follow-up; occurrence/recurrence of acute diverticulitis; need of surgery.

The study will take three year. The investigators aim at confirming that DICA classification is a valid parameter to predict the risk of acute diverticulitis occurrence/recurrence and the need of surgery in patients suffering from diverticulosis/diverticular disease of the colon. This could permit to select populations at higher or lower risk, having or not benefit from scheduled (and type) treatment able to reduce those risks.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopic diagnosis of diverticula in the colon

Exclusion Criteria:

* • Radiological signs (by abdominal CT or by ultrasounds) of acute diverticulitis (complicated or uncomplicated)

  * Inflammatory bowel diseases;
  * Ischemic colitis;
  * Prior colonic resection
  * Patients with severe liver failure (Child-Pugh C);
  * Patients with severe kidney failure;
  * Pregnant women;
  * Women of childbearing potential not using a highly effective method of contraception;
  * Patients who are currently using or who have received any laxative agents < 2 weeks prior to the enrollment;
  * Patients who are currently using or who have received mesalamine compounds < 2 weeks prior to the enrollment;
  * Patients who are currently using or who have received any probiotic agents < 2 weeks prior to the enrollment;
  * Nonsteroidal anti-inflammatory drug (NSAID) use < 1 week prior to the enrollment;
  * Patients who have received treatment with antibiotics (even those not absorbed) < 2 weeks prior to the enrollment;
  * Inability to comply with study protocol and to give informed consensus to the procedure;
  * Patients with or history of cancer, of any origin, within 5 years before enrollment
  * History of alcohol, drug, or chemical abuse
  * Any severe pathological condition that may interfere with the proper study execution.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients accessing the endoscopic service
Sampling Method: Non-Probability Sample
Enrollment: 2215 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
DICA score and diverticulitis | 3 years
  Correlation between appearance of diverticulitis and DICA score.

SECONDARY OUTCOMES:
DICA score and surgery | 3 years
  Correlation between need to colonic surgery for complicated diverticular disease and DICA score.
DICA score and therapy | 3 years
  Correlation between response to treatment and DICA score.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Tursi, MD, Principal Investigator — Gastroenterology Service , ASL BAT, Andria (BT) - Italy; Giovanni Brandimarte, MD, Study Director — UOC di Medicina Interna, Servizio di Endoscopia Digestiva, Ospedale "Cristo Re" Rome; Walter Elisei, MD, Principal Investigator — UOC di Gastroenterologia, ASL Roma 6 Albano Laziale (Rome); Marcello Picchio, MD, Principal Investigator — UOC di Chirurgia Generale, Ospedale "P. Colombo", ASL Roma 6 Velletri (Rome)
Locations (45):
- Brazil (2):
  - Av, 470 - Hosp Ort de Goiania (St Aeroporto), Goiânia, Goiás
  - Consultório R, 46 - 25 Clin de Gastroentero, Goiânia, Goiás
- Italy (38):
  - UOC di Gastroenterologia, Ospedale "San Pio da Pietrelcina", Vasto, Chieti
  - Sapienza University of Rome- Polo Pontino, Terracina, Latina
  - UOC di Gastroenterologia, Ospedale "Santa Caterina Novella", Galatina, Lecce
  - Servizio Gastroenterologia ed Endoscopia Digestiva, Casa di Cura "Villa dei Pini", Civitanova Marche, Macerata
  - IBD Unit, Ospedale Universitario "Humanitas", Rozzano, Milan
  - UOC di Gastroenterologia, Policlinico "San Donato", San Donato Milanese, Milan
  - UO di Endoscopia Digestiva, Nuovo Ospedale Civile "Sant'Agostino Estense", Baggiovara, Modena
  - UOC di Gastroenterologia, Ospedale "T. Maresca", Torre del Greco, Napoli
  - SS di Endoscopia Digestiva, Ospedale "San Matteo degli Infermi" Spoleto (PG), Spoleto, Perugia
  - Servizio di Gastroenterologia ed Endoscopia Digestiva, Casa della Salute Magliano Sabina, Magliano Sabina, Rieti
  - UOC di Gastroenterologia, ASL Roma 6, Albano Laziale, Roma
  - UOC di Gastroenterologia ed Endoscopia Chirurgica, Ospedale "Grassi", Ostia Antica, Rome
  - UOC di Chirurgia Generale, Ospedale "P. Colombo", ASL Roma 6, Velletri, Rome
  - SSD di Endoscopia Digestiva, Ospedale "Valle d'Itria, Martina Franca, Taranto
  - UO Endoscopia Digestiva, ULSS4 Alto Vicentino,, Santorso, Vicenza
  - UOSD di Endoscopia Digestiva, Ospedale di Tarquinia, Tarquinia, Viterbo
  - Gastroenterology Service , ASL BAT,, Andria
  - Sezione di Medicina Interna, Clinica Medica "A. Murri", Policlinico Consorziale, Bari
  - UOC di Gastroenterologia, Ospedale "San Paolo", Bari
  - UO di Gastroenterologia - Policlinico del Monserrato, Università di Cagliari, Cagliari
  - UOC di Gastroenterologia, Ospedale "Pugliese-Ciaccio", Catanzaro
  - U.O.D. di Endoscopia Digestiva, Ospedale "S. Maria Goretti", Latina
  - UOC di Gastroenterologia, Ospedale "San Salvatore", Università de L'Aquila L'Aquila, L’Aquila
  - UOC di Gastroenterologia, A.O. "L. Sacco" , Università di Milano, Milan
  - UOS di Gastroenterologia ed Endoscopia Digestiva- Ospedale "Bucchieri - La Ferla", Palermo
  - UO di Gastroenterologia - Ospedale Maggiore, Università di Parma, Parma
  - Dipartimento di medicina Clinica e Sperimentale, Sezione di Gastroenterologia ed Epatologia Ospedale "Santa Maria della Misericordia" Hospital, Università di Perugia,, Perugia
  - SC di Gastroenterologia - Endoscopia Digestiva, IRCCS Arcispedale "Santa Maria Nuova", Reggio Emilia
  - UOD di Endoscopia Digestiva e Nutrizionale, Ospedale "S. Eugenio", Rome
  - UOC di Chirurgia Generale "I", Policlinico "Umberto I", Università "Sapienza", Rome
  - UOC di Medicina Interna, Servizio di Endoscopia Digestiva, Ospedale "Cristo Re" Roma, Rome
  - UOC di Medicina Interna e Gastroenterologia, C.I. "Columbus", Università Cattolica, Rome
  - UOC di Medicina Interna e Gastroenterologia, Policlinico "A. Gemelli", Rome
  - UOC di Gastroenterologia ed Endoscopia Digestiva, A.O. "S. Giovanni-Addolorata", Rome
  - Servizio di Gastroenterologia ed Endoscopia Digestiva, PTP "Nuovo Regina Margherita", Rome
  - UOC di Gastroenterologia, Ospedale "Molinette", Turin
  - UOC di Gastroenterologia, Ospedale "Santa Maria della Misericordia", Udine
  - UOC di Gastroenterologia, Ospedale "Belcolle", Viterbo
- Centre for abdominal surgery, Vilnius University Hospital Santariskiu Klinikos,, Vilnius, Lithuania
- Department of Gastroenterology, Hepatology and Clinical Oncology, Medical Postgraduate Education Centre; Department of Gastrointestinal Oncology, Maria Sklodowska-Curie Clinical Oncology Institute, Warsaw, Poland
- 2nd Medical Department, Iuliu Hatieganu University of Medicine and Pharmacy, Cluj-Napoca, Cluj, Romania
- Department of Colorectal Surgery, Kings College Hospital,, London, United Kingdom
- Universidad Central de Venezuela, Loira Medical Center,, Caracas, Venezuela

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tursi A, Brandimarte G, Di Mario F, Andreoli A, Annunziata ML, Astegiano M, Bianco MA, Buri L, Cammarota G, Capezzuto E, Chilovi F, Cianci M, Conigliaro R, Del Favero G, Di Cesare L, Di Fonzo M, Elisei W, Faggiani R, Farroni F, Forti G, Germana B, Giorgetti GM, Giovannone M, Lecca PG, Loperfido S, Marmo R, Morucci P, Occhigrossi G, Penna A, Rossi AF, Spadaccini A, Zampaletta C, Zilli M, Zullo A, Scarpignato C, Picchio M. Development and validation of an endoscopic classification of diverticular disease of the colon: the DICA classification. Dig Dis. 2015;33(1):68-76. doi: 10.1159/000366039. Epub 2014 Dec 17. PMID 25531499
- [Derived] Tursi A, Brandimarte G, Di Mario F, Elisei W, Picchio M, Allegretta L, Annunziata ML, Bafutto M, Bassotti G, Bianco MA, Colucci R, Conigliaro R, Dumitrascu D, Escalante R, Ferrini L, Forti G, Franceschi M, Graziani MG, Lammert F, Latella G, Maconi G, Nardone G, Camara de Castro Oliveira L, Chaves Oliveira E, Papa A, Papagrigoriadis S, Pietrzak A, Pontone S, Poskus T, Pranzo G, Reichert MC, Rodino S, Regula J, Scaccianoce G, Scaldaferri F, Vassallo R, Zampaletta C, Zullo A, Piovani D, Bonovas S, Danese S; DICA International Group. Prognostic performance of the 'DICA' endoscopic classification and the 'CODA' score in predicting clinical outcomes of diverticular disease: an international, multicentre, prospective cohort study. Gut. 2022 Jul;71(7):1350-1358. doi: 10.1136/gutjnl-2021-325574. Epub 2021 Oct 26. PMID 34702716